CLINICAL TRIAL: NCT03126968
Title: Prophylactic Topical Epinephrine to Reduce Transbronchial Lung Biopsy-related Hemorrhage in Lung Transplant Recipients: a Prospective Double-blind Placebo-controlled Trial (PROPHylactic Epinephrine in Transbronchial Biopsy [PROPHET] Trial)
Brief Title: Prophylactic Topical Epinephrine to Reduce Bleeding in Transbronchial Lung Biopsies
Acronym: PROPHET
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Robert M Reed, Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HP-00070208
Record Dates: First submitted 2017-04-17; First posted 2017-04-25 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Lung Transplant; Complications, Mechanical; Lung Transplant; Complications; Bleeding; Hemoptysis
MeSH Terms: conditions — Hemorrhage; Hemoptysis | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prophylactic topical epinephrine (Experimental): Study participants who meet inclusion and exclusion criteria and allocated to this arm will be randomized to receive prophylactic endobronchial topical epinephrine in a blinded manner prior to performance of transbronchial lung biopsy.
  Interventions: Drug: Topical epinephrine
- Placebo (Placebo Comparator): Study participants who meet inclusion and exclusion criteria and allocated to this arm will be randomized to receive prophylactic endobronchial topical placebo in the form of normal saline in a blinded manner prior to performance of transbronchial lung biopsy.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Topical epinephrine — Prophylactic topical epinephrine
  Arms: Prophylactic topical epinephrine
Drug: Placebos — Topical placebo (normal saline)
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Bleeding poses potential for significant complication after transbronchial lung biopsies. The investigators hypothesize that prophylactic intrabronchial instillation of topical epinephrine will reduce the likelihood of bleeding. The investigators plan a double-blind, placebo controlled trial to evaluate this hypothesis.

DETAILED DESCRIPTION:
The role of prophylactic topical epinephrine in improving hemostasis and prevention of clinically-significant pulmonary hemorrhage has never been studied formally in the past, despite its common use by pulmonologists performing bronchoscopic TBLB. Lung transplant recipients undergo multiple bronchoscopies and TBLBs for surveillance and evaluation of ACR as well as lung infection, especially during the first year post-transplantation. This population may have a predilection to TBLB-related bleeding and may benefit from measures to reduce the frequency and magnitude of this relatively common complication.

In the PROPHET trial, the investigators intend to assess the degree of biopsy-related bleeding, measures taken to control bleeding, and potential effects of bleeding on completion of the intended procedure in 50 bronchoscopy procedures performed on single and double lung transplant recipients, randomized to prophylactic topical epinephrine versus placebo (normal saline). The study participant, physician performing the TBLB, and independent observer reviewing the procedure recording will all be blinded to the randomization. Further use of measures to control bleeding that occurs during the procedure as well as the decision to complete the procedure as planned or to abort it prematurely will be left to the discretion of the performer. In this way, the investigators aim to elucidate a potential role of topical epinephrine in the prevention of TBLB-related airway bleeding in lung transplant recipients and assess whether the dose and volume of instillation used in the investigators' institution comprises an effective means to prevent hemorrhagic complications of TBLB.

HYPOTHESIS

The investigators hypothesize that prophylactic instillation of topical epinephrine prior to performance of TBLB will decrease the frequency and extent of biopsy-related hemorrhage as well as result in fewer procedures being aborted earlier than intended due to bleeding complications as well as shorter overall procedure time due to the preventive effect on bleeding. Concomitantly, the investigators hypothesize that the instillation of topical epinephrine will not be associated with a serious adverse event profile in comparison to placebo.

SPECIFIC AIMS

In this randomized-controlled double blind placebo controlled clinical trial post-lung transplant patients scheduled to receive bronchoscopy with TBLB as part of their routine standard of care will be randomized to receive a fixed dose and volume of topical endobronchial epinephrine versus matching volume of placebo which will be instilled into the target biopsy airway prior to performance of TBLB. This study will specifically aim at providing the following information:

Aim 1: Demonstrate the feasibility of assessments of bleeding related to TBLB, including:

1. The degree of TBLB-related bleeding using a standardized grading scale used by the physician performing the procedure to quantify the degree of procedure-related bleeding.
2. The degree of TBLB-related bleeding using a standardized grading scale used by two independent observers blinded to patient data and study drug assignment who will review a video recording of the procedure to quantify the degree of procedure-related bleeding.
3. The magnitude of inter-observer variability in grading TBLB-related hemorrhage based on review of video recording of the procedure.

Aim 2: Evaluate the hypothesis that prophylactic administration of topical epinephrine results in reductions in TBLB-related hemorrhage in lung transplant recipients, including:

1. The frequency of active measures taken to control pulmonary hemorrhage once it occurred.
2. The proportion of procedures completed as planned in terms of obtaining a predefined target number of biopsy specimens.
3. Comparison between single- and double-lung transplant recipients in terms of prevalence and degree of TBLB-related hemorrhage.
4. Identification of clinical factors associated with an increased or decreased risk of procedure-related hemorrhage.

Aim 3: Evaluate the hypothesis that prophylactic administration of topical epinephrine affects the overall efficiency of bronchoscopy with TBLB performance, including:

1. Overall duration of the bronchoscopic procedure.
2. The proportion of procedures completed as planned in terms of number of adequate biopsies obtained as assessed by the physician performing the bronchoscopy.
3. The proportion of procedures resulting in acquisition of adequate biopsy samples that allows proper pathologic evaluation of assignment of a pathologic diagnosis.

Aim 4: Explore the hypothesis that instillation of our prespecified dose and volume of topical epinephrine into the target biopsy airway is not associated with an adverse event profile that is significantly different from placebo, including:

1. The prevalence of clinically significant hemodynamic changes.
2. The prevalence of cardiac adverse events, including conduction abnormalities, arrhythmia, and myocardial ischemia.
3. The prevalence of other vascular adverse events, including stroke, mesenteric ischemia, and critical limb ischemia.
4. Identification of clinical factors associated with an increased or decreased risk of drug-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ≥18 years of age.
* Single- or double-lung transplant recipients scheduled for bronchoscopy with TBLB.
* Willingness to sign an informed consent for study participation.

Exclusion Criteria:

* Age <18 years.
* Pregnancy.
* Inability to understand and provide a written informed consent.

Exclusion criteria for TBLB:

* Platelet count <50 K/microL.
* International normalized ratio (INR) >1.5.
* Known bleeding diathesis.
* Use of prophylactic or therapeutic dose of unfractionated heparin within 6 hours of the procedure.
* Use of prophylactic dose of low molecular weight heparin within 12 hours of the procedure.
* Use of therapeutic dose of low molecular weight heparin within 24 hours of the procedure.
* Use of oral direct thrombin inhibitors or oral factor 10a inhibitors within 48 hours of the procedure.
* Use of clopidogrel, ticlopidine, ticagrelor, or prasugrel within 5 days of the procedure.
* Uremia, defined as estimated glomerular filtration rate (eGFR) ≤30 mL/min.
* Moderate to severe pulmonary hypertension as defined by a mean pulmonary artery pressure of >40 mm Hg on right heart catheterization or an estimated pulmonary artery systolic pressure of >62 mm Hg on transthoracic echocardiography, both performed within 1 year of the procedure.
* An additional synchronous procedure with possible bleeding (bronchoalveolar lavage and endobronchial biopsy allowed).
* Decompensated liver cirrhosis, defined as the presence of clinically significant ascites, clinical evidence of esophageal or gastric varices, or history of bleeding from gastric or esophageal varices.
* Prior history of TBLB-related airway bleeding requiring admission to the hospital or advanced measures to achieve hemostasis, including endotracheal intubation, bronchial blocker application, bronchial artery embolization, or surgical intervention.

Exclusion criteria for application of topical epinephrine:

* Systolic heart failure with an ejection fraction (EF) of <35% as assess by echocardiography performed within one year prior to the procedure.
* Myocardial infarction, acute coronary syndrome, percutaneous coronary intervention, or coronary artery bypass surgery within 6 months prior to the procedure.
* Symptoms and/or ECG findings suggestive of ongoing cardiac ischemia on the day of the procedure.
* Moderate- to severe-grade cardiac valvulopathy as assessed by echocardiography performed within one year prior to the procedure.
* Inadequately controlled supraventricular arrhythmia, including atrial fibrillation, atrial flutter, and atrio-ventricular node re-entrant tachycardia (AVNRT) as revealed by ECG or cardiac monitoring at the time of the procedure.
* Presence of an internal cardioverter/defibrillator.
* History of second or third degree (complete) heart block or sick sinus syndrome.
* Baseline ECG or cardiac monitoring revealing frequent occurrence (≥10 events per minute) of atrial or ventricular ectopy documented prior to or at the time of the procedure.
* History of ventricular arrhythmias requiring pharmacologic or electrical cardioversion within the 2 years preceding the procedure.
* Serum potassium of <3.0 mmol/L within the week prior to the procedure.
* Serum glucose level of ≥300 mg/dL within the week prior to the procedure.
* Any history of critical ischemia related to peripheral arterial disease.
* Persistent resting heart rate (HR) measurement of ≥120 beats per minute prior to or at the time of the procedure.
* Persistent resting systolic blood pressure (SBP) measurement of ≥180 mm Hg prior to or at the time of the procedure.
* Persistent resting diastolic blood pressure (DBP) measurement of ≥110 mm Hg prior to or at the time of the procedure.
* History of acute closed-angle glaucoma within one year of the procedure.
* Diagnosis of pheochromocytoma requiring pharmacologic therapy with an alpha adrenoreceptor blocker at the time of the procedure.
* Diagnosis of thyrotoxicosis requiring pharmacologic therapy with an anti-thyroid agent at the time of the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Reed, MD, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - University of Maryland Medical Center - Midtown Campus, Baltimore, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen HA, Fontana RS, Sanderson DR, Harrison EG Jr. Transbronchoscopic lung biopsy in diffuse pulmonary disease: results in 300 cases. Med Clin North Am. 1970 Jul;54(4):951-9. No abstract available. PMID 5425117
- [Background] Fletcher EC, Levin DC. Flexible fiberoptic bronchoscopy and fluoroscopically guided transbronchial biopsy in the management of solitary pulmonary nodules. West J Med. 1982 Jun;136(6):477-83. PMID 7113195
- [Background] Prakash UB, Offord KP, Stubbs SE. Bronchoscopy in North America: the ACCP survey. Chest. 1991 Dec;100(6):1668-75. doi: 10.1378/chest.100.6.1668. PMID 1959412
- [Background] Ahmad M, Livingston DR, Golish JA, Mehta AC, Wiedemann HP. The safety of outpatient transbronchial biopsy. Chest. 1986 Sep;90(3):403-5. doi: 10.1378/chest.90.3.403. PMID 3743154
- [Background] Hernandez Blasco L, Sanchez Hernandez IM, Villena Garrido V, de Miguel Poch E, Nunez Delgado M, Alfaro Abreu J. Safety of the transbronchial biopsy in outpatients. Chest. 1991 Mar;99(3):562-5. doi: 10.1378/chest.99.3.562. PMID 1995209
- [Background] Leslie KO, Gruden JF, Parish JM, Scholand MB. Transbronchial biopsy interpretation in the patient with diffuse parenchymal lung disease. Arch Pathol Lab Med. 2007 Mar;131(3):407-23. doi: 10.5858/2007-131-407-TBIITP. PMID 17516743
- [Background] Berbescu EA, Katzenstein AL, Snow JL, Zisman DA. Transbronchial biopsy in usual interstitial pneumonia. Chest. 2006 May;129(5):1126-31. doi: 10.1378/chest.129.5.1126. PMID 16685001
- [Background] Poletti V, Ravaglia C, Buccioli M, Tantalocco P, Piciucchi S, Dubini A, Carloni A, Chilosi M, Tomassetti S. Idiopathic pulmonary fibrosis: diagnosis and prognostic evaluation. Respiration. 2013;86(1):5-12. doi: 10.1159/000353580. Epub 2013 Jun 26. PMID 23816667
- [Background] Matthay RA, Farmer WC, Odero D. Diagnostic fibreoptic bronchoscopy in the immunocompromised host with pulmonary infiltrates. Thorax. 1977 Oct;32(5):539-45. doi: 10.1136/thx.32.5.539. PMID 594932
- [Background] Cazzadori A, Di Perri G, Todeschini G, Luzzati R, Boschiero L, Perona G, Concia E. Transbronchial biopsy in the diagnosis of pulmonary infiltrates in immunocompromised patients. Chest. 1995 Jan;107(1):101-6. doi: 10.1378/chest.107.1.101. PMID 7813258
- [Background] Gilman MJ, Wang KP. Transbronchial lung biopsy in sarcoidosis. An approach to determine the optimal number of biopsies. Am Rev Respir Dis. 1980 Nov;122(5):721-4. doi: 10.1164/arrd.1980.122.5.721. PMID 7447156
- [Background] Pinsker KL, Kamholz SL. Diagnosis of sarcoidosis by transbronchial lung biopsy. Chest. 1981 Jan;79(1):123-4. doi: 10.1378/chest.79.1.123b. No abstract available. PMID 7449494
- [Background] Talmage EA. Safe combined general and topical anesthesia for laryngoscopy and bronchoscopy. South Med J. 1973 Apr;66(4):455-9. doi: 10.1097/00007611-197304000-00015. No abstract available. PMID 4575235
- [Background] Kukafka DS, O'Brien GM, Furukawa S, Criner GJ. Surveillance bronchoscopy in lung transplant recipients. Chest. 1997 Feb;111(2):377-81. doi: 10.1378/chest.111.2.377. PMID 9041985
- [Background] Papin TA, Lynch JP 3rd, Weg JG. Transbronchial biopsy in the thrombocytopenic patient. Chest. 1985 Oct;88(4):549-52. doi: 10.1378/chest.88.4.549. PMID 4042705
- [Background] Jain P, Sandur S, Meli Y, Arroliga AC, Stoller JK, Mehta AC. Role of flexible bronchoscopy in immunocompromised patients with lung infiltrates. Chest. 2004 Feb;125(2):712-22. doi: 10.1378/chest.125.2.712. PMID 14769756
- [Background] Jabbardarjani H, Eslaminejad A, Mohammadtaheri Z, Kiani A, Arab A, Masjedi MR. The effect of cup versus alligator forceps on the results of transbronchial lung biopsy. J Bronchology Interv Pulmonol. 2010 Apr;17(2):117-21. doi: 10.1097/LBR.0b013e3181dc9920. PMID 23168725
- [Background] Sehgal IS, Bal A, Dhooria S, Agrawal P, Gupta N, Ram B, Aggarwal AN, Behera D, Agarwal R. A Prospective Randomized Controlled Trial Comparing the Efficacy and Safety of Cup vs Alligator Forceps for Performing Transbronchial Lung Biopsy in Patients With Sarcoidosis. Chest. 2016 Jun;149(6):1584-6. doi: 10.1016/j.chest.2016.03.025. No abstract available. PMID 27287583
- [Background] Flick MR, Wasson K, Dunn LJ, Block AJ. Fatal pulmonary hemorrhage after transbronchial lung biopsy through the fiberoptic bronchoscope. Am Rev Respir Dis. 1975 Jun;111(6):853-6. doi: 10.1164/arrd.1975.111.6.853. PMID 1137250
- [Background] Chhajed PN, Aboyoun C, Malouf MA, Hopkins PM, Plit ML, Glanville AR. Risk factors and management of bleeding associated with transbronchial lung biopsy in lung transplant recipients. J Heart Lung Transplant. 2003 Feb;22(2):195-7. doi: 10.1016/s1053-2498(02)00462-x. PMID 12581769
- [Background] Zavala DC. Diagnostic fiberoptic bronchoscopy: Techniques and results of biopsy in 600 patients. Chest. 1975 Jul;68(1):12-9. doi: 10.1378/chest.68.1.12. PMID 168036
- [Background] Glanville AR. The role of surveillance bronchoscopy post-lung transplantation. Semin Respir Crit Care Med. 2013 Jun;34(3):414-20. doi: 10.1055/s-0033-1348466. Epub 2013 Jul 2. PMID 23821514
- [Background] Sahebjami H. Letter: Iced saline lavage during bronchoscopy. Chest. 1976 Jan;69(1):131-2. doi: 10.1378/chest.69.1.131b. No abstract available. PMID 1244274
- [Background] Du Rand IA, Blaikley J, Booton R, Chaudhuri N, Gupta V, Khalid S, Mandal S, Martin J, Mills J, Navani N, Rahman NM, Wrightson JM, Munavvar M; British Thoracic Society Bronchoscopy Guideline Group. British Thoracic Society guideline for diagnostic flexible bronchoscopy in adults: accredited by NICE. Thorax. 2013 Aug;68 Suppl 1:i1-i44. doi: 10.1136/thoraxjnl-2013-203618. No abstract available. PMID 23860341
- [Background] Lee P, Mehta AC, Mathur PN. Management of complications from diagnostic and interventional bronchoscopy. Respirology. 2009 Sep;14(7):940-53. doi: 10.1111/j.1440-1843.2009.01617.x. PMID 19740256
- [Background] Solomonov A, Fruchter O, Zuckerman T, Brenner B, Yigla M. Pulmonary hemorrhage: A novel mode of therapy. Respir Med. 2009 Aug;103(8):1196-200. doi: 10.1016/j.rmed.2009.02.004. Epub 2009 Feb 28. PMID 19251406
- [Background] Marquez-Martin E, Vergara DG, Martin-Juan J, Flacon AR, Lopez-Campos JL, Rodriguez-Panadero F. Endobronchial administration of tranexamic Acid for controlling pulmonary bleeding: a pilot study. J Bronchology Interv Pulmonol. 2010 Apr;17(2):122-5. doi: 10.1097/LBR.0b013e3181dc8c17. PMID 23168726
- [Background] Shigemura N, Wan IY, Yu SC, Wong RH, Hsin MK, Thung HK, Lee TW, Wan S, Underwood MJ, Yim AP. Multidisciplinary management of life-threatening massive hemoptysis: a 10-year experience. Ann Thorac Surg. 2009 Mar;87(3):849-53. doi: 10.1016/j.athoracsur.2008.11.010. PMID 19231404
- [Background] Yendamuri S. Massive Airway Hemorrhage. Thorac Surg Clin. 2015 Aug;25(3):255-60. doi: 10.1016/j.thorsurg.2015.04.009. Epub 2015 Jun 12. PMID 26210922
- [Background] Aboyoun CL, Tamm M, Chhajed PN, Hopkins P, Malouf MA, Rainer S, Glanville AR. Diagnostic value of follow-up transbronchial lung biopsy after lung rejection. Am J Respir Crit Care Med. 2001 Aug 1;164(3):460-3. doi: 10.1164/ajrccm.164.3.2011152. PMID 11500350
- [Background] Vitulo P, Cremaschi P, Arbustini E, Volpato G, Volpini E, Martinelli L, Fracchia C, Rossi A. Surveillance transbronchial biopsy in the diagnosis of acute lung rejection in heart and lung and lung transplant recipients. Monaldi Arch Chest Dis. 1996 Feb;51(1):12-5. PMID 8901314
- [Background] Trulock EP, Ettinger NA, Brunt EM, Pasque MK, Kaiser LR, Cooper JD. The role of transbronchial lung biopsy in the treatment of lung transplant recipients. An analysis of 200 consecutive procedures. Chest. 1992 Oct;102(4):1049-54. doi: 10.1378/chest.102.4.1049. PMID 1327662
- [Background] Baz MA, Layish DT, Govert JA, Howell DN, Lawrence CM, Davis RD, Tapson VF. Diagnostic yield of bronchoscopies after isolated lung transplantation. Chest. 1996 Jul;110(1):84-8. doi: 10.1378/chest.110.1.84. PMID 8681672
- [Background] Timofte I, Terrin M, Barr E, Sanchez P, Kim J, Reed R, Britt E, Ravichandran B, Rajagopal K, Griffith B, Pham S, Pierson RN 3rd, Iacono A. Belatacept for renal rescue in lung transplant patients. Transpl Int. 2016 Apr;29(4):453-63. doi: 10.1111/tri.12731. Epub 2016 Feb 8. PMID 26678245
- [Background] Chan CC, Abi-Saleh WJ, Arroliga AC, Stillwell PC, Kirby TJ, Gordon SM, Petras RE, Mehta AC. Diagnostic yield and therapeutic impact of flexible bronchoscopy in lung transplant recipients. J Heart Lung Transplant. 1996 Feb;15(2):196-205. PMID 8672524
- [Background] Inoue M, Minami M, Wada N, Nakagiri T, Funaki S, Kawamura T, Shintani Y, Okumura M. Results of surveillance bronchoscopy after cadaveric lung transplantation: a Japanese single-institution study. Transplant Proc. 2014 Apr;46(3):944-7. doi: 10.1016/j.transproceed.2013.10.055. PMID 24767387
- [Background] GOGERTY JH, STRAND HA, OGILVIE AL, DILLE JM. Vasopressor effects of topical epinephrine in certain dental procedures. Oral Surg Oral Med Oral Pathol. 1957 Jun;10(6):614-22. doi: 10.1016/s0030-4220(57)80009-7. No abstract available. PMID 13441276
- [Background] Zamani A. Bronchoscopic intratumoral injection of tranexamic acid: a new technique for control of biopsy-induced bleeding. Blood Coagul Fibrinolysis. 2011 Jul;22(5):440-2. doi: 10.1097/MBC.0b013e328346efb7. PMID 21577092
- [Background] Zamani A. Bronchoscopic intratumoral injection of tranexamic acid to prevent excessive bleeding during multiple forceps biopsies of lesions with a high risk of bleeding: a prospective case series. BMC Cancer. 2014 Mar 1;14:143. doi: 10.1186/1471-2407-14-143. PMID 24581173
- [Background] Higgins TS, Hwang PH, Kingdom TT, Orlandi RR, Stammberger H, Han JK. Systematic review of topical vasoconstrictors in endoscopic sinus surgery. Laryngoscope. 2011 Feb;121(2):422-32. doi: 10.1002/lary.21286. Epub 2011 Jan 13. PMID 21271600
- [Background] Valdes CJ, Bogado M, Rammal A, Samaha M, Tewfik MA. Topical cocaine vs adrenaline in endoscopic sinus surgery: a blinded randomized controlled study. Int Forum Allergy Rhinol. 2014 Aug;4(8):646-50. doi: 10.1002/alr.21325. Epub 2014 Mar 26. PMID 24678064
- [Background] Fernandez-Cossio S, Rodriguez-Dinten MJ, Gude F, Fernandez-Alvarez JM. Topical Vasoconstrictors in Cosmetic Rhinoplasty: Comparative Evaluation of Cocaine Versus Epinephrine Solutions. Aesthetic Plast Surg. 2016 Oct;40(5):637-44. doi: 10.1007/s00266-016-0673-2. Epub 2016 Jun 29. PMID 27357633
- [Background] Korkmaz H, Yao WC, Korkmaz M, Bleier BS. Safety and efficacy of concentrated topical epinephrine use in endoscopic endonasal surgery. Int Forum Allergy Rhinol. 2015 Dec;5(12):1118-23. doi: 10.1002/alr.21590. Epub 2015 Jul 8. PMID 26152362
- [Background] Orlandi RR, Warrier S, Sato S, Han JK. Concentrated topical epinephrine is safe in endoscopic sinus surgery. Am J Rhinol Allergy. 2010 Mar-Apr;24(2):140-2. doi: 10.2500/ajra.2010.24.3454. PMID 20338114
- [Background] Papp AA, Uusaro AV, Ruokonen ET. The effects of topical epinephrine on haemodynamics and markers of tissue perfusion in burned and non-burned patients requiring skin grafting. Burns. 2009 Sep;35(6):832-9. doi: 10.1016/j.burns.2008.10.001. Epub 2009 May 30. PMID 19481869
- [Background] Kuster GG, Fischer B. Pharmacologic hemostasis in laparoscopy: topical epinephrine facilitates cholecystectomy. Am Surg. 1993 May;59(5):281-4. PMID 8489094
- [Background] Roberts JR, Greenberg MI, Knaub MA, Kendrick ZV, Baskin SI. Blood levels following intravenous and endotracheal epinephrine administration. JACEP. 1979 Feb;8(2):53-6. doi: 10.1016/s0361-1124(79)80036-2. PMID 439542
- [Background] Mazkereth R, Paret G, Ezra D, Aviner S, Peleg E, Rosenthal T, Barzilay Z. Epinephrine blood concentrations after peripheral bronchial versus endotracheal administration of epinephrine in dogs. Crit Care Med. 1992 Nov;20(11):1582-7. doi: 10.1097/00003246-199211000-00017. PMID 1424703
- [Background] Mall W, Abel H. Topical application of epinephrine during bronchoscopy in barbiturate-halothane-anaesthesia and its influence on cardiac action. Bronchopneumologie. 1978 Jul-Aug;28(4):311-6. PMID 92354
- [Background] Janjua M, Badshah A, Allen SA. Images in cardiology. Epinephrine-induced ST elevation: a case of endobronchial topical epinephrine-induced coronary vasospasm. Heart. 2009 Apr;95(8):656. doi: 10.1136/hrt.2008.161646. No abstract available. PMID 19329720
- [Background] Steinfort DP, Herth FJ, Eberhardt R, Irving LB. Potentially fatal arrhythmia complicating endobronchial epinephrine for control of iatrogenic bleeding. Am J Respir Crit Care Med. 2012 May 1;185(9):1028-30. doi: 10.1164/ajrccm.185.9.1028. No abstract available. PMID 22550217
- [Background] Khoo KL, Lee P, Mehta AC. Endobronchial epinephrine: confusion is in the air. Am J Respir Crit Care Med. 2013 May 15;187(10):1137-8. doi: 10.1164/rccm.201209-1682LE. No abstract available. PMID 23675717
- [Background] Steinfort DP, Herth FJ, Eberhardt R, Irving LB. Reply: Endobronchial epinephrine: confusion is in the air. Am J Respir Crit Care Med. 2013 May 15;187(10):1138. doi: 10.1164/rccm.201301-0123LE. No abstract available. PMID 23675719
- [Background] Paret G, Vaknin Z, Ezra D, Peleg E, Rosenthal T, Vardi A, Mayan H, Barzilay Z. Epinephrine pharmacokinetics and pharmacodynamics following endotracheal administration in dogs: the role of volume of diluent. Resuscitation. 1997 Aug;35(1):77-82. doi: 10.1016/s0300-9572(96)01091-x. PMID 9259064
- [Background] Diette GB, Wiener CM, White P Jr. The higher risk of bleeding in lung transplant recipients from bronchoscopy is independent of traditional bleeding risks: results of a prospective cohort study. Chest. 1999 Feb;115(2):397-402. doi: 10.1378/chest.115.2.397. PMID 10027438
- [Background] Hopkins PM, Aboyoun CL, Chhajed PN, Malouf MA, Plit ML, Rainer SP, Glanville AR. Prospective analysis of 1,235 transbronchial lung biopsies in lung transplant recipients. J Heart Lung Transplant. 2002 Oct;21(10):1062-7. doi: 10.1016/s1053-2498(02)00442-4. PMID 12398870
- [Derived] Kalchiem-Dekel O, Tran BC, Glick DR, Ha NT, Iacono A, Pickering EM, Shah NG, Sperry MG, Sachdeva A, Reed RM. Prophylactic epinephrine attenuates severe bleeding in lung transplantation patients undergoing transbronchial lung biopsy: Results of the PROPHET randomized trial. J Heart Lung Transplant. 2023 Sep;42(9):1205-1213. doi: 10.1016/j.healun.2023.03.007. Epub 2023 Mar 14. PMID 37140517
- [Derived] Kalchiem-Dekel O, Iacono A, Pickering EM, Sachdeva A, Shah NG, Sperry M, Tran BC, Reed RM. Prophylactic epinephrine for the prevention of transbronchial lung biopsy-related bleeding in lung transplant recipients (PROPHET) study: a protocol for a multicentre randomised, double-blind, placebo-controlled trial. BMJ Open. 2019 Mar 23;9(3):e024521. doi: 10.1136/bmjopen-2018-024521. PMID 30904852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients undergoing bronchoscopy with transbronchial biopsies after lung transplantation were offered participation in the study.
Pre-assignment Details: Patients not meeting eligibility criteria were not included. Informed consent was obtained immediately prior to the procedure. Patients were randomized in a double-blind, placebo-controlled fashion.
Units Other Than Participants: Procedures
Period: Overall Study
Arm/Group | Prophylactic Topical Epinephrine | Placebo
Started | 33; 46 Procedures | 33; 54 Procedures
Completed | 33; 46 Procedures | 33; 54 Procedures
Not Completed | 0; 0 Procedures | 0; 0 Procedures

BASELINE CHARACTERISTICS:
Population: Study consisted of 100 procedures performed on 66 participants as participants were permitted to participate more than once.
Units Other Than Participants: Procedures
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylactic Topical Epinephrine | Placebo | Total
Number analyzed (Participants) | 33 | 33 | 66
Number analyzed (Procedures) | 46 | 54 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [55 to 68] | 64 [56 to 68] | 63.5 [56 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 22 | 21 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race / Ethnicity: African American | 10 | 12 | 22
  Race / Ethnicity: Latino | 1 | 4 | 5
  Race / Ethnicity: Caucasian | 22 | 17 | 39

OUTCOME MEASURES:

1. Primary Outcome: Intra-procedural Hemorrhage Grading by the Performing Bronchoscopist
Description: Intra-procedural hemorrhage will be graded by the performing bronchoscopist according to the following scale:
  1. No hemorrhage.
  2. Mild hemorrhage - Any bleeding originating from the biopsy target airway requiring wedging of the bronchoscope or "in and out" motion in order to achieve hemostasis.
  3. Moderate hemorrhage - Any bleeding originating from the biopsy target airway requiring in addition to maneuvering the bronchoscope application of iced saline or topical epinephrine or placing the patient with the bleeding lung in the dependent position.
  4. Severe hemorrhage - Any bleeding originating from the biopsy target airway requiring, in addition to the above-mentioned maneuvers, early termination of the procedure or necessitating application of balloon tamponade, endotracheal intubation, application of a bronchial blocker, or use of other invasive measures to achieve hemostasis, such as bronchial artery embolization or surgical intervention.
Time Frame: This outcome will be analyzed at the time of procedure performance and up to 48 hours following the procedure.
Measure: Count of Units; unit: Procedures
Units Other Than Participants: Procedures
Arm/Group | Prophylactic Topical Epinephrine | Placebo
Number analyzed (Participants) | 33 | 33
Number analyzed (Procedures) | 46 | 54
Procedures
  Severe or very severe hemorrhage | 4 | 13
  Moderate, severe, or very severe hemorrhage | 11 | 24
  Unblinded administration of epinephrine for bleeding | 8 | 20
  Early termination of the procedure due to bleeding | 4 | 13

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Prophylactic Topical Epinephrine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 4/33 | 4/33
Other Adverse Events (participants affected / at risk) | 16/33 | 18/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylactic Topical Epinephrine (N=33) | Placebo (N=33)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) — Iatrogenic pneumothorx
Hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) — Deterioration requiring escalation of care (admission to hospital in both cases)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylactic Topical Epinephrine (N=33) | Placebo (N=33)
Drop in BP >20 from baseline (Cardiac disorders) | 16 (16) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT03126968/Prot_SAP_002.pdf